CLINICAL TRIAL: NCT05671562
Title: A Randomised Placebo-controlled Trial to Investigate the Effect of Lactolycopene on Sperm Quality in Men With a Low Total Motile Sperm Count: a Pilot Study.
Brief Title: The Effect of Lycopene on Sperm Quality in Men Attending Fertility Clinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: Health Education England, Wessex (Other); Manchester Metropolitan University (Other); University of Sheffield (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: STH22299
Record Dates: First submitted 2022-12-15; First posted 2023-01-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Total Motile Sperm Count
MeSH Terms: interventions — Lycopene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lycopene (Experimental): Capsules containing 7mg of lycopene. 2 capsules are swallowed once per day with water for 12 weeks. Looks identical to placebo capsule.
  Interventions: Dietary Supplement: Lycopene
- Placebo (Placebo Comparator): Placebo capsules containing an inactive ingredient. 2 capsules are swallowed once per day with water for 12 weeks. Looks identical to lycopene capsule.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lycopene — Capsule containing lycopene 7mg x 2 daily for 12 weeks
  Arms: Lycopene
Dietary Supplement: Placebo — Capsule containing inactive substance 7mg x 2 daily for 12 weeks
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to test whether lycopene (an antioxidant found in cooked tomatoes) will improve the number of swimming sperm in the ejaculates of men with low total motile sperm count.

Participants will take either lycopene capsules or identical capsules containing no lycopene for 12 weeks. We will analyse the quality of their semen before and after taking the capsules, and compare the results.

Hypothesis: Supplementation with lycopene will improve testicular function (semen quality) in males with low total motile sperm count (TMSC).

DETAILED DESCRIPTION:
Impaired testicular function contributes to around 50% of heterosexual infertility and is often characterized by a low total motile sperm count. Evidence suggests that one cause of low total motile sperm count is oxidative stress within the ejaculate, where harmful oxygen species damage the sperm. Antioxidants to combat oxidative stress within the ejaculate have been proposed as a method of increasing the total motile sperm count. Lycopene is a powerful antioxidant found abundantly in cooked tomatoes and has been shown to improve testicular function in a healthy population. This double blinded randomised controlled trial aims to investigate whether lycopene can improve testicular output in participants with a low motile sperm count. Semen analysis will be carried out before and after the intervention. The intervention is a commercially available lycopene capsule or an identical placebo.

Hypothesis: Supplementation with lactolycopene will improve testicular function (semen quality) in males with low total motile sperm count (TMSC).

ELIGIBILITY:
Inclusion Criteria:

1. Males aged 18 - 50 years of age
2. Attending the Fertility Clinic at the Jessop Wing, (Sheffield Teaching Hospitals).
3. Found to have poor testicular function as evidenced by a low motile sperm count (<20 million motile sperm per ejaculate).
4. Willing to comply with the study procedures and provide informed consent.

Exclusion Criteria:

1. Participants who report allergy to tomatoes, whey, soy.
2. Men with previous testicular surgery or a current or previous diagnosis of cancer.
3. Men found to have normal sperm parameters.
4. Known infection with hepatitis or HIV.
5. Men with azoospermia

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2023-05-03 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Total motile sperm count | Change from Baseline total motile sperm count at 12 weeks
  Number of swimming sperm in the total ejaculate

SECONDARY OUTCOMES:
Sperm motility | Change from Baseline sperm motility at 12 weeks
  % of swimming sperm
Sperm concentration | Change from Baseline sperm concentration at 12 weeks
  Number of sperm per ml of ejaculate
Sperm morphology | Change from Baseline sperm morphology at 12 weeks
  Appearance of sperm
Sperm DNA fragmentation | Change from Baseline sperm DNA fragmentation at 12 weeks
  % of sperm with fragmented DNA
Oxidative reductive potential of semen | Change from Baseline semen oxidative reductive potential at 12 weeks
  To compare level of oxidants and antioxidants within the sample

CONTACTS AND LOCATIONS:
Overall Officials: Lucy Wood, Principal Investigator — National Health Service, United Kingdom
Locations (1):
- Jessop Fertility, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No